CLINICAL TRIAL: NCT04699071
Title: Phase II Trial of Lenvatinib Plus PembrolizumAb in Recurrent Gynecological Clear Cell Adenocarcinomas (LARA)
Brief Title: Trial of Lenvatinib Plus PembrolizumAb in Recurrent Gynecological Clear Cell Adenocarcinomas (LARA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY01/05/20
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinomas; Recurrent Gynecological
Keywords: Lenvatinib; PembrolizumAb; gynecological; Adenocarcinomas
MeSH Terms: conditions — Adenocarcinoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: combination therapy of continuous daily oral lenvatinib with three-weekly intravenous pembrolizumab in patients with recurrent clear cell carcinoma of gynecological origin (CCGC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with recurrent clear cell carcinoma of gynecological origin (CCGC) (Experimental): Recurrent clear cell carcinoma of gynecological origin (ovarian and endometrial primary) after progression on chemotherapy.
  Interventions: Drug: pembrolizumab and lenvatinib

INTERVENTIONS:
Drug: pembrolizumab and lenvatinib — All patients will receive oral lenvatinib daily plus intravenous pembrolizumab 3-weekly.
  A cycle is 21 days. Allowances will be made for stepwise dose reductions of lenvatinib due to treatment-related toxicities.
  Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, (CTCAE) Version 5.0.
  Patients are planned to continue therapy until disease progression, intolerable toxicity, or withdrawal of patient consent.

SUMMARY:
This is a phase II non-randomized, multi-center study. The primary end point of this study is the objective response rate (ORR) at 24 weeks, using response evaluation criteria for solid tumors (RECIST) 1.1 criteria, for the combination therapy of continuous daily oral lenvatinib with three-weekly intravenous pembrolizumab in patients with recurrent clear cell carcinoma of gynecological origin (CCGC). The statistical design is Simon's minimax two-stage design and the present study aims to complete stage 1 of the Simon's two-stage design.

DETAILED DESCRIPTION:
Primary Objective

(1) Objective: To determine the efficacy as measured by the objective response rate (ORR) at 24 weeks using RECIST 1.1 criteria when patients with recurrent CCGCs are treated with lenvatinib plus pembrolizumab.

Hypothesis: The ORR (complete response plus partial response) at 24 weeks seen in recurrent CCGC patients treated with lenvatinib plus pembrolizumab combination therapy will be improved compared to historical control (hypothesized ORR of 30% with combination therapy compared to historical ORR of ORR of 10% with chemotherapy).

Primary Endpoint: The ORR at 24 weeks using RECIST 1.1 criteria when patients with recurrent CCGCs are treated with lenvatinib plus pembrolizumab.

Secondary Objectives,

1. Objective: To determine the efficacy of lenvatinib plus pembrolizumab in recurrent CCGCs.

   Hypothesis: The ORR by immune RECIST (iRECIST) criteria, progression-free survival (PFS) rate and clinical benefit rate (CBR) (complete response plus partial response plus stable disease) at 24 weeks, as well as duration of response and PFS observed in recurrent CCGC patients treated with lenvatinib plus pembrolizumab combination therapy will be improved compared to historical control.

   Endpoint: To determine the ORR using iRECIST criteria at 24 weeks when patients with recurrent CCGCs are treated with lenvatinib plus pembrolizumab.

   Endpoint: To assess the duration of response when patients with recurrent CCGCs are treated with lenvatinib plus pembrolizumab.

   Endpoint: To assess the PFS when patients with recurrent CCGCs are treated with lenvatinib plus pembrolizumab.

   Endpoint: To determine the 24 week PFS rate of lenvatinib plus pembrolizumab in this population.

   Endpoint: To determine the CBR at 24 weeks of lenvatinib plus pembrolizumab in this population.
2. Objective: To describe the adverse event (AE) profile of lenvatinib plus pembrolizumab in this patient population.

Exploratory Objectives

1. Clinical Objectives: To evaluate the effect of potential prognostic factors (baseline patient and tumor characteristics, notably: initial performance status, stage at diagnosis and platinum-free interval), on the efficacy of lenvatinib plus pembrolizumab in this population.
2. Translational Objectives: To evaluate the pre- to post-treatment changes in the frequency of tumor-associated macrophages (TAMs) in patients receiving lenvatinib plus pembrolizumab.
3. Translational Objectives: To evaluate the pre- to post-treatment changes in the frequency and gene expression profile of different lymphocyte (e.g. CD4, CD8, Treg, B cells) and myeloid (e.g. DCs, MDSCs) subsets in patients receiving lenvatinib plus pembrolizumab.
4. Translational Objectives: To identify predictive biomarkers of response in patients receiving lenvatinib plus pembrolizumab (e.g. PD-1/PD-L1/VEGF expression).
5. Translational Objectives: To evaluate the pre-to post-treatment changes in the concentration of relevant cytokines/chemokines (e.g.: GM-CSF, G-CSF, VEGFA, IL2, IL12, IL13, IL6, Interferons) in patients receiving lenvatinib plus pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of recurrent CCGC (ovarian and endometrial primary), as evidenced by WT-1 negativity, will be enrolled in this study. For tumors with a mixed histology, at least 70% of the tumor must consist of clear cell carcinoma.

  2. Patients must have had at least one prior line of platinum-based chemotherapy in the course of their treatment paradigm. A maximum of 4 prior lines of systemic treatment regimens will be allowed and may include chemotherapy and biologics (prior immune checkpoint inhibitor treatment will not be permitted).

  3. Participants must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment.

  4. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
  1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
  2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.

     5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

     6. Have at least 1 measurable lesion based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

     7. Provision of an archived tumor tissue block (or at least 10 newly cut unstained slides) where such samples exist in a quantity sufficient to allow for analysis.

     8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.

     9. Life expectancy exceeding 12 weeks.

     10. Have adequate organ function as defined in the following. Specimens must be collected within 10 days prior to the start of study treatment.

     Haematology i) Absolute neutrophil count (ANC) ≥1500/µL ii) Platelets ≥100 000/µL iii) Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La

     Renal I) Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR

     ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

     Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

     Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

     Exclusion Criteria:
* 1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

  2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).

  3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing. The safety of resumption of lenvatinib after resolution of wound healing has not been established".

  4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.

  5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

  6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

  7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

  8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.

  9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.

  10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

  11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.

  12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.

  13. Has an active infection requiring systemic therapy.

  14. Has a known history of Human Immunodeficiency Virus (HIV) infection.

  15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detectable HCV RNA) infection.

  16. Has a known history of active TB (Bacillus Tuberculosis).

  17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

  18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

  19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

  20. Has had an allogenic tissue/solid organ transplant.

  21. Has uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.

  22. Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.

  23. Has known bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.

  24. Has > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 4 years
  the percentage of subjects with a confirmed CR or PR as per RECIST 1.1 criteria.
Progression-free survival | 4 years
  time from enrolment to the first documented tumor progression, or death due to any cause whichever occurred first. PFS time of any living patient with no documented progression, or any patient starting other cytotoxic and/or cytostatic therapies, will be censored at the date of last evaluable disease assessment on-study. PFS time of patients with no evaluable disease assessment on-study will be censored at enrollment
Duration of response | 4 years
  This will be measured from the time measurement criteria for CR/PR (whichever is first recorded) are first met until the first date that recurrent or progressive disease is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: David Shao Peng Tan, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] del Carmen MG, Birrer M, Schorge JO. Clear cell carcinoma of the ovary: a review of the literature. Gynecol Oncol. 2012 Sep;126(3):481-90. doi: 10.1016/j.ygyno.2012.04.021. Epub 2012 Apr 21. PMID 22525820
- [Result] Brinton LA, Felix AS, McMeekin DS, Creasman WT, Sherman ME, Mutch D, Cohn DE, Walker JL, Moore RG, Downs LS, Soslow RA, Zaino R. Etiologic heterogeneity in endometrial cancer: evidence from a Gynecologic Oncology Group trial. Gynecol Oncol. 2013 May;129(2):277-84. doi: 10.1016/j.ygyno.2013.02.023. Epub 2013 Feb 26. PMID 23485770
- [Derived] Ngoi NYL, Lee JY, Lim D, Thian YL, Lim YW, Chan JJ, Chay WY, Zhang Z, Gopinathan A, Lim SE, Low J, Ng J, Tong P, Lee YJ, Park J, Kim JW, Tan TZ, Zhu J, Tai BC, Choi CH, Kim BG, Tan DSP. Pembrolizumab plus lenvatinib in recurrent gynaecological clear cell carcinoma (LARA): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2026 Jan 15:S1470-2045(25)00662-X. doi: 10.1016/S1470-2045(25)00662-X. Online ahead of print. PMID 41548565